CLINICAL TRIAL: NCT07304635
Title: Comparison of Postoperative Analgesic Effectiveness of Erector Spinae Plane Block and Combined With Superficial Parasternal Intercostal Plane Block Within the Enhanced Recovery After Cardiac Surgery (ERACS) Program: A Prospective, Randomized, Double-Blind Study
Brief Title: Comparison of the Postoperative Analgesic Effectiveness of Erector Spinae Plane Block Versus Its Combination With Superficial Parasternal Intercostal Plane Block Within the ERACS Program
Acronym: ERACS-ESP-SPIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, FATMA CANDAN YEREBAKAN, Principal Investigator, Ankara University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ERACSDEL001
Record Dates: First submitted 2025-12-12; First posted 2025-12-26 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-10

CONDITIONS: Sternotomy; Postoperative Delirium; Postoperative Pain Management
Keywords: sternotomy; post-sternotomy pain; postoperative pain; postoperative delirium; erector spinae plane blocks; superficial parasternal intercostal plane blocks
MeSH Terms: conditions — Emergence Delirium; Pain, Postoperative | interventions — Parapsychology; Dental Occlusion

STUDY DESIGN:
Intervention Model Description: This study is designed as a prospective, randomized, double-blind, parallel-group clinical trial conducted within the Enhanced Recovery After Cardiac Surgery (ERACS) program.
  A total of 42 adult patients undergoing elective cardiac surgery via median sternotomy will be randomized in a 1:1 ratio into two groups using a computer-generated randomization sequence and sealed opaque envelopes.
  Group E: Bilateral erector spinae plane (ESP) block
  Group EP: Bilateral ESP block combined with superficial parasternal intercostal plane (SPIP) block
  Both interventions will be performed under ultrasound guidance after induction of general anesthesia.
  Postoperative assessments-including VAS pain scores, sedation (RASS), and delirium screening (Nu-DESC)-will be recorded at standardized time points up to 72 hours after extubation.
  The study aims to compare postoperative analgesic effectiveness and the impact of pain control on postoperative delirium.
Who Masked: Participant, Investigator
Masking Description: The study will be double-blind, meaning neither the researchers nor the participants will know which treatment group they belong to, ensuring unbiased outcome assessment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: Erector Spinae Plane Block (Group E) (Experimental): After induction of general anesthesia, patients will receive a bilateral ultrasound-guided erector spinae plane block at the T4--T5 vertebral level.
  A total of 30 mL of 0.25% bupivacaine per side (prepared as 10 mL saline + 10 mL 0.5% bupivacaine per syringe) will be injected into the deep fascial plane beneath the erector spinae muscle using an 80 mm block needle under aseptic conditions.
  The spread of the local anesthetic will be observed in a craniocaudal direction in real time. The procedure will be repeated bilaterally.
  All patients will subsequently receive standardized postoperative analgesia with paracetamol 1 g IV every 6 hours; if VAS > 4, tramadol 50 mg IV will be given as rescue analgesia.
  Interventions: Procedure: Procedure: Erector Spinae Plane (ESP) Block
- Erector Spinae Plane Block + Superficial Parasternal Intercostal Plane Block (Group EP) (Active Comparator): Following induction of general anesthesia, patients will receive a bilateral ESP block (same technique as in Group E) with 20 mL of 0.25% bupivacaine per side.
  Afterward, a bilateral superficial parasternal intercostal plane block (SPIP) will be performed in the 4th-5th intercostal spaces, approximately 2-3 cm lateral to the midline, using a linear ultrasound probe and 80 mm block needle.
  After confirming negative aspiration and hydrodissection with 1-3 mL saline, 10 mL of 0.25% bupivacaine per side will be injected into the interfacial plane.
  The total local anesthetic volume for both blocks combined will be 60 mL, kept below the toxic threshold.
  Standard postoperative analgesia will be identical to Group E (paracetamol 1 g IV every 6 hours, and tramadol 50 mg IV if VAS > 4).
  Interventions: Procedure: Erector Spinae Plane (ESP) Block + Superficial Parasternal Intercostal Plane (SPIP) Block

INTERVENTIONS:
Procedure: Procedure: Erector Spinae Plane (ESP) Block — A bilateral ultrasound-guided erector spinae plane block will be performed at the T4-T5 vertebral level after induction of general anesthesia.
  Using an 80 mm peripheral nerve block needle and an in-plane approach, 30 mL of 0.25% bupivacaine per side will be injected into the fascial plane deep to the erector spinae muscle.
  The spread of the local anesthetic will be visualized in real time in a craniocaudal direction.
  This technique provides multidermatomal somatic and visceral analgesia (approximately T2-T9).
  Arms: Arm 1: Erector Spinae Plane Block (Group E)
Procedure: Erector Spinae Plane (ESP) Block + Superficial Parasternal Intercostal Plane (SPIP) Block — After induction of general anesthesia, patients will receive:
  Bilateral ESP block with 20 mL of 0.25% bupivacaine per side, performed as described above at the T5 level, and
  Bilateral SPIP block performed at the 4th-5th intercostal spaces, approximately 2-3 cm lateral to the midline, using a linear ultrasound probe.
  For the SPIP block, after confirming needle placement with hydrodissection (1-3 mL saline) and negative aspiration, 10 mL of 0.25% bupivacaine per side will be injected between the pectoralis major and external intercostal muscles.
  Arms: Erector Spinae Plane Block + Superficial Parasternal Intercostal Plane Block (Group EP)

SUMMARY:
This prospective, randomized, double-blind, parallel-group clinical trial within the Enhanced Recovery After Cardiac Surgery (ERACS) program compares postoperative analgesic effectiveness of bilateral erector spinae plane (ESP) block versus ESP combined with superficial parasternal intercostal plane (SPIP) block in adult patients undergoing elective cardiac surgery via median sternotomy.

DETAILED DESCRIPTION:
Rationale: Effective multimodal, opioid-sparing analgesia is crucial in cardiac surgery to enhance recovery and reduce pulmonary and cognitive complications. Neuraxial techniques (e.g., epidural) carry increased hematoma risk under anticoagulation; hence, fascial plane blocks like ESP and SPIP are safer alternatives.

Methodology: Randomized (ResearchRandomizer.org), 1:1 allocation, opaque sealed envelopes. ESP and SPIP performed under ultrasound guidance at standardized doses and locations.

Blinding: Patients and postoperative evaluators are blinded; block-performing anesthesiologist unblinded but uninvolved in assessment.

Follow-up: 0-72 hours after extubation with predefined time points for VAS, RASS, and Nu-DESC evaluations.

ELIGIBILITY:
Inclusion Criteria

* Patients scheduled for elective cardiac surgery via median sternotomy under the ERACS protocol
* Age between 18 and 80 years
* ASA physical status II-III
* Body Mass Index (BMI) between 18 and 35 kg/m²
* No cognitive impairment (able to cooperate and follow commands)
* No history of chronic pain or regular analgesic use
* Provided written informed consent after detailed explanation of the study

Exclusion Criteria

* Age < 18 years or > 80 years
* ASA physical status ≥ IV
* Emergency surgery
* Pregnant or breastfeeding women
* Redo coronary artery bypass surgery
* Pre-existing cognitive disorder or psychiatric illness affecting pain or delirium evaluation
* Infection or skin lesion at the injection site
* Known allergy or hypersensitivity to local anesthetics (bupivacaine or amide type)
* Chronic pain or opioid use prior to surgery
* Unwillingness to participate or withdrawal of consent at any stage

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2024-08-30 (Actual); Primary Completion 2025-07-27 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
VAS (resting) | Up to 72 hours post-extubation
  Average of VAS scores at 0, 1, 6, 12, 24, 48, and 72 hours after extubation (t=0). Lower scores indicate better analgesia.
  Pain was assessed using the 0-10 Visual Analog Scale (VAS).
  Pain severity was classified as follows:
  0 = no pain, 1-3 = mild pain, 4-6 = moderate pain, 7-10 = severe pain. Rescue analgesia was administered when VAS score was > 4.

SECONDARY OUTCOMES:
VAS (movement) | 0-72 hours
  Mean VAS scores during movement at all time points
Total rescue tramadol use (mg) | 0-72 hours
  Cumulative IV tramadol dose
Time to first rescue analgesic (min) | 0-72 hours
  Time between extubation and first rescue tramadol
Delirium incidence (Nu-DESC ≥ 2) | 12, 24, 48, 72 hours
  Nursing Delirium Screening Scale (Nu-DESC) score ≥ 2 Delirium was assessed using the Nursing Delirium Screening Scale (NU-DESC). NU-DESC consists of five items, each scored from 0 to 2 (total score: 0-10). A total NU-DESC score ≥ 2 was considered positive for delirium.
  Items:
  Disorientation Inappropriate behavior Inappropriate communication Illusions / hallucinations Psychomotor retardation
RASS score profile | 0, 12, 24, 48, 72 hours
  Richmond Agitation-Sedation Scale distribution Sedation level was assessed using the Richmond Agitation-Sedation Scale (RASS).
  RASS scores were classified as:
  * 4 = combative,
  * 3 = very agitated,
  * 2 = agitated,
  * 1 = restless, 0 = alert and calm,
    * 1 = drowsy,
    * 2 = light sedation,
    * 3 = moderate sedation,
    * 4 = deep sedation,
    * 5 = unarousable.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara University Faculty of Medicine, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No